CLINICAL TRIAL: NCT06396585
Title: The Efficacy and Safety of Tislelizumab Combined With Anlotinib and S1 Plus Oxaliplatin as Neoadjuvant Therapy for the Locally Advanced Adenocarcinoma of Esophagogastric Junction : a Prospective，Single-arm, Phase II Trial (TASTE Trial)
Brief Title: The Efficacy and Safety of Tislelizumab Combined With Anlotinib and S1 Plus Oxaliplatin as Neoadjuvant Therapy for the Locally Advanced Adenocarcinoma of Esophagogastric Junction
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TASTE Trial
Record Dates: First submitted 2024-04-30; First posted 2024-05-02 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Immunotherapy Gastroesophageal Junction
MeSH Terms: interventions — tislelizumab; anlotinib; Oxaliplatin; Tegafur

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab combined with anlotinib chemotherapy (Experimental)
  Interventions: Drug: Tislelizumab; Drug: Anlotinib; Drug: Oxaliplatin; Drug: Tegafur

INTERVENTIONS:
Drug: Tislelizumab — Participants will receive Tislelizumab, 200mg, intravenously over 30 - 60 minutes, day 1 ,Q3W
Drug: Anlotinib — Participants will receive anlotinib,12mg, qd，d1-d14，Q3W
Drug: Oxaliplatin — Participants will receive Oxaliplatin, 130mg/m2, iv, day 1 ,Q3W
Drug: Tegafur — Participants will receive S-1 40-60mg/m2/c次，bid ，d1-d14，Q3W

SUMMARY:
To evaluate the efficacy and safety of tislelizumab combined with antilotinib and SOX regimen for neoadjuvant treatment of locally advanced esophagogastric junction cancer

ELIGIBILITY:
Inclusion Criteria:

* Female and male patient ≥ 18 and ≤ 75 years.
* Histologically confirmed, medically operable, resectable adenocarcinoma of the gastroesophageal junction (AEG, Siewert II-III)，uT3, uT4a, uT4b any N category, M0, or any T N+ M0 patient
* ECOG≤1
* No previous surgical treatment, anti-tumor chemoradiotherapy/immunotherapy was performed.
* Exclusion of distant metastases by CT or MRI of abdomen, pelvis, and thorax, bone scan or MRI (if bone metastases are suspected due to clinical signs).
* Preoperative endoscopic examination confirmed no positive peritoneal implantation metastasis and exfoliated cells.
* The expected survival time is more than 6 months.
* Women of childbearing age shall be those who agree to use contraception (such as intrauterine devices, contraceptives or condoms) during the study and for 6 months after the end of the study; those who have a negative serum or urine pregnancy test within 7 days before study enrollment and must be non-lactating; and men who agree to use contraception during the study and for 6 months after the end of the study.
* Hematological, hepatic and renal function parameters adequate to allow surgical procedure and chemotherapy
* Patient able and willing to provide written informed consent and to comply with the study protocol and with the planned surgical procedures

Exclusion Criteria:

* Diagnosis of malignant diseases other than gastric cancer within 5 years prior to first administration (excluding radical basal cell carcinoma of the skin, squamous carcinoma of the skin, and/or radical resectable carcinoma in situ).
* Significant clinical bleeding symptoms or clear bleeding tendency, such as gastrointestinal bleeding, hemorrhagic gastric ulcer or vasculitis, etc. occurred within 3 months before enrollment. If fecal occult blood was positive at baseline, reexamination could be performed, if it was still positive after reexamination, gastroscopy was required.
* Prior treatment: anti-PD-1, anti-PD-L1, or anti-PD-L2 drugs or drugs that target another stimulating or co-inhibiting T-cell receptor (e.g., CTLA-4, OX-40, CD137).
* A history of immunodeficiency, including HIV testing positive.
* Is currently participating in an interventional clinical study or has been treated with another study drug or study device in the 4 weeks prior to initial dosing.
* Patients who had a history of cardiovascular and cerebrovascular diseases and were still taking thrombolytic drugs or anticoagulants orally.
* HER2 positive is known.
* Patients with previous gastrointestinal perforation, abdominal abscess or recent intestinal obstruction (within 3 months) or imaging or clinical symptoms suggesting intestinal obstruction.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response | 4 weeks after surgery
  Total tumor regression rate under pathologyPrimary tumor or lymph node surgery specimen pathological examination without residual tumor cell

SECONDARY OUTCOMES:
Major pathological response | 4 weeks after surgery
  Total/moderate tumor regression rate under pathologyPrimary tumor or lymph node surgery specimen pathological examination without residual tumor cell
Objective Response Rate (ORR) | At the end of Cycle 3 (each cycle is 21 days)
  Objective Response Rate Determine the tumor shrinkage rate, tumor boundary and the adhesion of tumor

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian cancer hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No